CLINICAL TRIAL: NCT00002752
Title: PHASE I STUDY OF ANTI-TENASCIN MONOCLONAL ANTIBODY 131I 81C6 VIA SURGICALLY CREATED CYSTIC RESECTION CAVITY IN THE TREATMENT OF PATIENTS WITH PRIMARY OR METASTATIC MALIGNANT BRAIN TUMORS
Brief Title: Radiolabeled Monoclonal Antibody Therapy in Treating Patients With Primary or Metastatic Brain Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: Pro00004635; DUMC-2426-01-2R8 (Other: DUMC); DUMC-000223-00-2R7 (Other: DUMC); DUMC-0328-99-2R6 (Other: DUMC); DUMC-221-96-2R3 (Other: DUMC); DUMC-307-97-2R4; DUMC-307-98-2R5; NCI-H96-0009; CDR0000064688 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2003-07-08 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2013-02

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer
Keywords: childhood supratentorial ependymoma; recurrent childhood brain tumor; recurrent adult brain tumor; adult medulloblastoma; adult glioblastoma; tumors metastatic to brain; childhood high-grade cerebral astrocytoma; adult anaplastic astrocytoma; adult myxopapillary ependymoma; adult anaplastic ependymoma; adult anaplastic oligodendroglioma; adult mixed glioma; adult pilocytic astrocytoma; adult subependymoma; adult ependymoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood medulloblastoma; newly diagnosed childhood ependymoma; recurrent childhood ependymoma; adult oligodendroglioma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Medulloblastoma; Glioblastoma; Astrocytoma; Ependymoma; Oligodendroglioma; Glioma; Glioma, Subependymal; Neuroectodermal Tumors, Primitive; Familial ependymoma; Gliosarcoma

INTERVENTIONS:
Radiation: iodine I 131 monoclonal antibody 81C6

SUMMARY:
RATIONALE: Radiolabeled monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of radiolabeled monoclonal antibody therapy in treating patients who have primary or metastatic brain cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects of intracranial iodine I 131 labeled anti-tenascin monoclonal antibody 81C6 in patients with primary or metastatic anaplastic gliomas.
* Determine the objective therapeutic response of these patients treated with this regimen.

OUTLINE: This is a dose escalation study of iodine I 131 labeled anti-tenascin monoclonal antibody 81C6 (MOAB 81C6). Patients are stratified by prior external beam radiotherapy (yes vs no).

Patients receive iodine I 131 labeled MOAB 81C6 intraventricularly followed by unlabeled MOAB 81C6 intraventricularly.

Cohorts of 3-6 patients receive escalating doses of iodine I 131 labeled MOAB 81C6 until the maximum tolerated dose is determined. The MTD is defined as the highest dose preceding that at which 3 of 6 patients experience dose-limiting toxicity.

Patients are followed monthly for 2 years, every 2 months for 2 years, and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 3-6 patients per cohort will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven primary or metastatic malignant supratentorial anaplastic glioma

  * Newly diagnosed or recurrent
  * No diffusely infiltrating or multifocal tumor
  * No tumor with subependymal spread
* Resection of glioma and placement of an intralesional catheter into the surgical cavity required before study
* Measurable lesion on enhanced CT scan or MRI

  * No measurable enhancing lesion greater than 1.0 cm beyond cavity margin
* Neoplastic cell reactivity with tenascin demonstrated by immunohistology with either a polyclonal rabbit antibody or a monoclonal murine antibody

PATIENT CHARACTERISTICS:

Age:

* 3 and over

Performance status:

* Karnofsky 50-100%

Hematopoietic:

* Absolute neutrophil count greater than 1,000/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 mg/dL
* AST less than 1.5 times normal
* Alkaline phosphatase less than 1.5 times normal

Renal:

* Creatinine less than 1.2 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 weeks since prior chemotherapy unless unequivocal evidence of tumor progression

Endocrine therapy:

* Corticosteroids allowed if at lowest possible dose and dose stable for at least 10 days prior to entry

Radiotherapy:

* At least 3 months since prior radiotherapy to site of measurable disease unless unequivocal evidence of tumor progression

Surgery:

* See Disease Characteristics

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1993-02; Primary Completion 2003-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke Cancer Institute
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States